CLINICAL TRIAL: NCT01997281
Title: The Effect of Dietary Fiber-enriched Cereals on Glycemic Control and Secretion of Gut Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-1307-133-508; 0620132990 (Other: SNUH Institutional Review Board)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2014-08

CONDITIONS: Diabetes Mellitus
Keywords: dietary fiber; diabetes mellitus; gut hormone
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DF-cereal (Experimental): * dietary fiber-enriched cereal is provided with milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount of cereal: 79 g (285.7 kcal) for dinner and breakfast, 38.5g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
  Interventions: Dietary Supplement: dietary fiber-enriched cereal
- conventional cereal (Other): * conventional cereal is provided with milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount of cereal: 80g (285.7 kcal) for dinner and breakfast, 40g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
  Interventions: Other: conventional cereal

INTERVENTIONS:
Dietary Supplement: dietary fiber-enriched cereal — * provided with 300 mL (150 mL at 10 p.m.) of milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount: 79g for dinner and breakfast, 38.5g for night snack (10 p.m.)
  * one serving of steamed egg is added for dinner and breakfast
  Arms: DF-cereal
Other: conventional cereal — * provided with 300 mL (150 mL at 10 p.m.) of milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount: 80 g for dinner and breakfast, 40 g for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
  Arms: conventional cereal

SUMMARY:
The aim of this study is to assess whether dietary fiber-enriched cereals effect on postprandial glucose levels and plasma glucagon-like peptide 1 (GLP-1) and/or glucose-dependent insulinotropic polypeptide (GIP) concentration in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Fifteen subjects with type 2 diabetes mellitus will be provided with study meals based on either dietary fiber-enriched cereals or conventional cereals upon two separate admissions in a cross-over fashion. The study meals will be provided at 6 p.m. and 10 p.m. on the day of admission, and 8 a.m. on the next day. A hamburger with coke as mixed meal will be given for lunch at noon on the second day. Blood sampling will be done every 30 minutes from 8 a.m. to 4 p.m. on the second day. The plasma levels of glucose, GLP-1, GIP, insulin, glucagon, and free fatty acid will be measured.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* HbA1c 6.5~8.5%
* on life style modification or metformin monotherapy at the time of screening

Exclusion Criteria:

* on sulfonylurea or insulin therapy at the time of screening
* allergy to wheat, flour, other cereals or nuts
* lactose intolerance
* pregnancy / lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Study Chair — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim EK, Oh TJ, Kim LK, Cho YM. Improving Effect of the Acute Administration of Dietary Fiber-Enriched Cereals on Blood Glucose Levels and Gut Hormone Secretion. J Korean Med Sci. 2016 Feb;31(2):222-30. doi: 10.3346/jkms.2016.31.2.222. Epub 2016 Jan 26. PMID 26839476

RESULTS

PARTICIPANT FLOW:
Groups:
- DF-cereal, Then Conventional Cereal: * Dietary fiber-enriched cereal was provided with 300 mL of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 79g (285.7 kcal) for dinner and breakfast, 38.5g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg was added for dinner and breakfast
  after 1 week of wash-out period, subjects were re-admitted
  * Conventional cereal was provided with 300 ml of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 80g (285.7 kcal) for dinner and breakfast, 40g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg wass added for dinner and breakfast
- Conventional Cereal, Then DF-cereal: * Conventional cereal was provided with 300 ml of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 80g (285.7 kcal) for dinner and breakfast, 40g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg wass added for dinner and breakfast
  after 1 week of wash-out period, subjects were re-admitted
  * Dietary fiber-enriched cereal was provided with 300 mL of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 79g (285.7 kcal) for dinner and breakfast, 38.5g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg was added for dinner and breakfast
Period: Overall Study
Arm/Group | DF-cereal, Then Conventional Cereal | Conventional Cereal, Then DF-cereal
Started | 7 | 7
Withdrawal | 1 | 0
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DF-cereal, Then Conventional Cereal | Conventional Cereal, Then DF-cereal | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.0) | 55.2 (8.0) | 55.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  South Korea | 6 | 7 | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.2 (2.0) | 25.0 (3.7) | 23.7 (2.9)
HbA1c [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 6.9 (0.7) | 6.7 (0.3) | 6.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Plasma Total GLP-1 Levels After Intake of the Study Meal
Description: To see the changes in the secretion of GLP-1 with dietary fiber enriched cereal, we will calculate the AUC of the plasma total GLP-1 levels.
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Measure: Mean (Standard Deviation); unit: pM x hr/L
Groups:
- DF-cereal: * dietary fiber-enriched cereal is provided with milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount of cereal: 79 g (285.7 kcal) for dinner and breakfast, 38.5g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
  dietary fiber-enriched cereal: - provided with 300 mL (150 mL at 10 p.m.) of milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount: 79g for dinner and breakfast, 38.5g for night snack (10 p.m.)
  * one serving of steamed egg is added for dinner and breakfast
- Conventional Cereal: * conventional cereal is provided with milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount of cereal: 80g (285.7 kcal) for dinner and breakfast, 40g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
  conventional cereal: - provided with 300 mL (150 mL at 10 p.m.) of milk, total 3 times (day 1: 6 p.m. and 10 p.m., day 2: 8 a.m.)
  * amount: 80 g for dinner and breakfast, 40 g for night snack (10 p.m.)
  * one serving (40g) of steamed egg is added for dinner and breakfast
Arm/Group | DF-cereal | Conventional Cereal
Number analyzed (Participants) | 13 | 13
pM x hr/L | 10.5 (1.9) | 10.5 (1.6)

2. Secondary Outcome: AUC of Plasma Total GIP Levels After Intake of the Study Meal
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Reporting Status: Not Posted

3. Secondary Outcome: AUC of Plasma Glucose Levels After Intake of the Study Meal
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Reporting Status: Not Posted

4. Secondary Outcome: AUC of Plasma Insulin Levels After Intake of the Study Meal
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Reporting Status: Not Posted

5. Secondary Outcome: AUC of Plasma Glucagon Levels After Intake of the Study Meal
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Reporting Status: Not Posted

6. Secondary Outcome: AUC of Serum Free Fatty Acid Levels After Intake of the Study Meal
Time Frame: every 30 minutes from 8 a.m. to noon on the second day
Reporting Status: Not Posted

7. Secondary Outcome: AUC of Plasma Total GIP Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

8. Secondary Outcome: AUC of Plasma Glucose Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

9. Secondary Outcome: AUC of Plasma Insulin Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

10. Secondary Outcome: AUC of Plasma Glucagon Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

11. Secondary Outcome: AUC of Serum Free Fatty Acid Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

12. Secondary Outcome: AUC of Plasma Total GLP-1 Levels After Lunch
Time Frame: every 30 minutes from noon to 4 p.m. on the second day
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The definition of adverse event and serious adverse event was not differ from clinicaltrials.gov definitions.
Groups:
- DF-cereal: * Dietary fiber-enriched cereal was provided with 300 mL of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 79g (285.7 kcal) for dinner and breakfast, 38.5g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg was added for dinner and breakfast
- Conventional Cereal: * Conventional cereal was provided with 300 ml of milk, total 3 times (Day 1 at 6 p.m. and 10 p.m., Day 2 at 8 a.m.)
  * amount of cereal: 80g (285.7 kcal) for dinner and breakfast, 40g (142.9 kcal) for night snack (10 p.m.)
  * one serving (40g) of steamed egg wass added for dinner and breakfast
Arm/Group | DF-cereal | Conventional Cereal
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 7/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DF-cereal (N=13) | Conventional Cereal (N=13)
abdominal discomfort (Gastrointestinal disorders) | 4 | 0
increased gas-out (Gastrointestinal disorders) | 2 | 0
increased amount and number of defecation (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes